CLINICAL TRIAL: NCT06600646
Title: Investigating the Role of ATP Production by Airway Epithelium in Patients With Refractory and Unexplained Chronic Cough (RCC/UCC).
Acronym: APEC
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: Hireb:17668
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Chronic Cough (CC)
Keywords: chronic cough; ATP; airway nerves
MeSH Terms: conditions — Chronic Cough | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bronchial Biopsies for RNA sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Refractory or Unexplained Chronic Cough
  Interventions: Diagnostic Test: Bronchoscopy
- Healthy Controls
  Interventions: Diagnostic Test: Bronchoscopy

INTERVENTIONS:
Diagnostic Test: Bronchoscopy — Bronchoscopy will be performed in patients with refractory or unexplained chronic cough and healthy controls.

SUMMARY:
Chronic cough is a common troublesome symptom which has a global prevalence of approximately 10%, but with wide variations across continents. Patients with refractory and unexplained chronic cough (RCC/UCC) often exhibit dysregulated vagal pathways, necessitating a neuronal biomarker for targeted treatment. ATP, involved in the ATP/P2X3 pathway, may serve as a potential biomarker due to its role in the cough reflex. The study aims to discover if ATP production by the airway epithelium is greater in RCC/UCC patients compared with healthy controls, if the epithelium is a source of ATP, whether gene and protein expression related to ATP production differs between these groups and whether ATP release is triggered by mechanical and chemical stimulation. Additionally, the study seeks to determine if biomarker gene expression signatures can differentiate RCC/UCC patients from healthy controls.

ELIGIBILITY:
Inclusion Criteria for RCC/UCC:

* Patients with a history of RCC/UCC.
* Normal Chest X-ray in the last 5 years.
* No Evidence of Airflow Obstruction (FEV1/FVC ratio above LLN)
* Cough Severity VAS ≥ 40 mm at screening.

Inclusion Criteria for Healthy Controls:

* No history of chronic cough, asthma, COPD, or clinical history of bronchiectasis or interstitial lung disease
* No current smokers or those with >10 pack year history.
* No evidence of airflow obstruction ( FEV1/FVC ratio above LLN).
* Able to understand and give written informed consent.

Exclusion Criteria:

* Participants who are currently established on treatment and their chronic cough is well controlled.
* Unable to perform acceptable and reproducible spirometry.
* Participants with a positive covid-19 test within 2 weeks of screening.
* Current smoker or ex-smoker with ≥20 pack year smoking history and abstinence of ≤6 months
* Symptoms of upper respiratory tract infection in the last 1 month which have not resolved
* Lower respiratory tract infection or pneumonia in the last 1 month
* Asthma exacerbation in the previous month requiring an increase or start of an inhaled corticosteroid (ICS) or oral corticosteroid (OCS)
* Significant other primary pulmonary disorders in particular; pulmonary embolism, pulmonary hypertension, lung cancer, cystic fibrosis, significant radiologically proven emphysema, interstitial lung disease or bronchiectasis.
* History of psychiatric illness, drug or alcohol abuse which may interfere in the participation of the trial.
* Allergy or intolerance to sedation medication including fentanyl and midazolam, or a history of complications during procedural sedation
* Severe coagulopathy, bleeding disorder, or medical need for anti- coagulation that would increase the risk of endobronchial biopsy as determined by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls will be recruited through local advertising, existing study databases or participation in previous studies where they have given permission to be contacted. Participants with RCC/UCC will be recruited by the investigators from existing study databases, clinics at either of the following sites:
  McMaster University Medical Centre, Department of Respiratory Medicine, 1200 Main St. West, Hamilton, Ontario, Canada, L8N 3Z5
  Firestone Institute for Respiratory Health, St Joseph's Healthcare, 50 Charlton Ave E, Hamilton, ON L8N 4A6
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in expressed genes | At baseline
  Expression of genes involved in intracellular ATP production, transport, extracellular metabolism in the airway epithelium will be compared in both RCC/UCC and healthy controls.

SECONDARY OUTCOMES:
Difference Immune Cells and Cytokines | 12 months
  Investigate differences in the levels of neuroinflammatory mediators and immune cells from the respiratory airways and distal alveoli.
Gene Expression | At baseline
  To compare the differences in RCC/UCC and healthy control in gene expression profiling in bronchial biopsies (sub-epithelial dominant).
Difference in Nerve Morphology | baseline
  Investigate differences in nerve length, nerve branch points, nerves expressive P2X3 receptors on airway sensory nerves expressing P2X3 receptor in RCC/UCC compared with healthy controls.
Difference in ATP release | 5,15,30 minutes
  ATP release from the cultured bronchial epithelial cells (BEC) taken from RCC/UCC and healthy controls after exposure to dynamic mechanical stretch and environmental exposures (cigarette smoke and NO2).

CONTACTS AND LOCATIONS:
Overall Officials: Imran Satia, MB BChir (cantab) MRCP PhD, Principal Investigator — McMaster University
Locations (1):
- Imran Satia, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This is an single visit of 15 patients with RCC/UCC compared with 15 Healthy Controls undergoing bronchoscopy at single centre in Hamilton, Ontario, Canada. Due to the small sample size individual level details will not be shared to protect confidentiality.